CLINICAL TRIAL: NCT04269954
Title: The Efficacy and Safety of Batroxobin Combined With Anticoagulation in Cerebral Venous Sinus Thrombosis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Ran Meng, Professor of neurology, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CVST2020
Record Dates: First submitted 2020-02-12; First posted 2020-02-17 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Cerebral Venous Sinus Thrombosis; Batroxobin
Keywords: Cerebral Venous Sinus Thrombosis
MeSH Terms: interventions — Heparin, Low-Molecular-Weight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Batroxobin combined with low molecular weight heparin (Experimental): Standard treatment of Batroxobin combined with low molecular weight heparin.
  Interventions: Drug: Batroxobin combined with low molecular weight heparin
- Low-molecular-weight heparin therapy (Other): Low-molecular-weight heparin combined with routine drug therapy.
  Interventions: Drug: Batroxobin combined with low molecular weight heparin

INTERVENTIONS:
Drug: Batroxobin combined with low molecular weight heparin — Standard treatment of Batroxobin combined with low molecular weight heparin

SUMMARY:
Our previous clinical case observations showed that batroxobin combined with anticoagulation therapy can improve the sinus recanalization rate in patients with CVST, shorten the hospital stay, and increase the neurological score of patients. Its main mechanism is to inhibit thrombosis after reducing fibrinogen, and to dissolve thrombus.

To further explore the safety of batroxobin combined with anticoagulation therapy for CVST, an open-label, randomized controlled (1: 1), single-center, prospective study was used. Further study on the safety and effectiveness of batroxobin combined with anticoagulation for CVST.

ELIGIBILITY:
Inclusion Criteria:

1. Cerebral venous thrombosis, confirmed by cerebral angiography (with intra-arterial contrast injection), magnetic resonance venography or computed tomographic venography.
2. Severe form of CVST with a high chance of incomplete recovery, as defined by the presence of one or more of the following risk factors

   1. Intracerebral hemorrhagic lesion due to CVST
   2. Mental status disorder
   3. Coma (Glasgow coma scale < 9)
   4. Thrombosis of the deep cerebral venous system
3. Uncertainty by the treating physician if ET or standard heparin therapy is the optimal therapy for the patient.

Exclusion Criteria:

1. Conditions associated with increased risk of bleeding
2. Any thrombolytic therapy within last 7 days
3. Cerebellar venous thrombosis with 4th ventricle compression and hydrocephalus, which requires surgery
4. Contraindication for anti-coagulant or batroxobin treatment 1)documented generalized bleeding disorder 2)concurrent thrombocytopenia (<100 x 10E9/L) 3)Fibrinogen below 100mg /dl 4)documented severe hepatic or renal dysfunction, that interferes with normal coagulation 5)uncontrolled severe hypertension (diastolic > 120 mm Hg) 6)known recent (< 3 months) gastrointestinal tract hemorrhage (not including hemorrhage from rectal hemorrhoids)
5. Any known associated condition (such as terminal cancer) with a poor short term (1 year) prognosis independent of CVST
6. Clinical and radiological signs of impending transtentorial herniation due to large space-occupying lesions (e.g. large cerebral venous infarcts or hemorrhages)
7. Recent (< 2 weeks) major surgical procedure (does not include lumbar puncture) or severe cranial trauma
8. Previously legally incompetent prior to CVST
9. Severe renal impairment
10. Active liver disease
11. Pregnancy, nursing or planning to become pregnant while in the trial
12. Further exclusion criteria apply
13. No informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With Major Bleeding Event (MBE) According to International Society on Thrombosis and Haemostasis (ISTH) Criteria in Full Observation Period | 2 weeks after randomization

SECONDARY OUTCOMES:
Favorable clinical outcome | 3 months after randomization
  modified Rankin score 0-1
Recanalization rate of cerebral venous system | 3 months after randomization
  DSA or MRV confirms cerebral venous sinus flow
Required surgical intervention in relation to CVST | 3 months after randomization
All cause mortality | 3 months after randomization

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Captial Medical University, Beijing, China

REFERENCES:
- [Result] Ding J, Zhou D, Hu Y, Elmadhoun O, Pan L, Ya J, Geng T, Wang Z, Ding Y, Ji X, Meng R. The efficacy and safety of Batroxobin in combination with anticoagulation on cerebral venous sinus thrombosis. J Thromb Thrombolysis. 2018 Oct;46(3):371-378. doi: 10.1007/s11239-018-1718-y. PMID 30062617
- [Result] Ding JY, Pan LQ, Hu YY, Rajah GB, Zhou D, Bai CB, Ya JY, Wang ZA, Jin KX, Guan JW, Ding YC, Ji XM, Meng R. Batroxobin in combination with anticoagulation may promote venous sinus recanalization in cerebral venous thrombosis: A real-world experience. CNS Neurosci Ther. 2019 May;25(5):638-646. doi: 10.1111/cns.13093. Epub 2019 Jan 23. PMID 30675757
- [Result] Yang Q, Duan J, Fan Z, Qu X, Xie Y, Nguyen C, Du X, Bi X, Li K, Ji X, Li D. Early Detection and Quantification of Cerebral Venous Thrombosis by Magnetic Resonance Black-Blood Thrombus Imaging. Stroke. 2016 Feb;47(2):404-9. doi: 10.1161/STROKEAHA.115.011369. Epub 2015 Dec 15. PMID 26670082